CLINICAL TRIAL: NCT01652274
Title: "Too Small for a Car Seat". An Unnoticed Obstacle to the Proper Use of Car Seats!
Brief Title: Level of Knowledge and Habitual Concepts of Turkish Parents on Child Passenger Safety
Status: Completed | Type: Observational
Sponsor: Fatih University (Other)
Responsible Party: Principal Investigator, Mehmet Kenan Kanburoglu, MD Kanburoglu, Fatih University
Other Study IDs: B 30 2 FTH 0 20 00 00/136; B 30 2 FTH 0 20 00 00/136 (Other: Fatih University Scientific Research Projects)
Record Dates: First submitted 2012-07-21; First posted 2012-07-30 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Equipment Safety; Accidents, Traffic
Keywords: Child Passenger Safety; Parental perception of vulnerability; Neonatology; Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mother: study objectives to Mother only
- Father: study objectives to Father only

SUMMARY:
It is well known that traffic accidents are one of the major reasons for death in childhood. Unfortunately scientific and statistical data usually comes from developed countries. In this study, the investigators will try to evaluate Turkish families' knowledge on Child Passenger Safety, observe how they carry their babies in the car and investigated the reasons behind the undesired behaviors.

ELIGIBILITY:
Inclusion Criteria:

* All families

Exclusion Criteria:

* Families with premature or neurologically disabled babies.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be done on mothers and fathers of babies brought to the first. control.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
test score | baseline
  test score that measures the level of knowledge on child passenger safety by a 10 item questionnaire

SECONDARY OUTCOMES:
Number of families using car seats properly | baseline
  I will be evaluated in 4 categories:
  Connecting the baby to the car seat properly, Connecting the car seat to the car properly, Using the rear facing, Placing the car seat to the center rear of the car.

OTHER OUTCOMES:
reasons for not using car seat | baseline
  face to face interview

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih University Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Committee on Injury, Violence, and Poison Prevention; Durbin DR. Child passenger safety. Pediatrics. 2011 Apr;127(4):788-93. doi: 10.1542/peds.2011-0213. Epub 2011 Mar 21. PMID 21422088
- [Background] Macy ML, Clark SJ, Freed GL, Butchart AT, Singer DC, Sasson C, Meurer WJ, Davis MM. Carpooling and booster seats: a national survey of parents. Pediatrics. 2012 Feb;129(2):290-8. doi: 10.1542/peds.2011-0575. Epub 2012 Jan 30. PMID 22291115
- [Background] Brown J, Hatfield J, Du W, Finch CF, Bilston LE. The characteristics of incorrect restraint use among children traveling in cars in New South Wales, Australia. Traffic Inj Prev. 2010 Aug;11(4):391-8. doi: 10.1080/15389588.2010.481770. PMID 20730686
- [Background] Dogan DG, Ertem IO, Karaaslan T, Forsyth BW. Perception of vulnerability among mothers of healthy infants in a middle-income country. Child Care Health Dev. 2009 Nov;35(6):868-72. doi: 10.1111/j.1365-2214.2009.01015.x. Epub 2009 Sep 4. PMID 19735267
- [Background] Bull MJ, Engle WA; Committee on Injury, Violence, and Poison Prevention and Committee on Fetus and Newborn; American Academy of Pediatrics. Safe transportation of preterm and low birth weight infants at hospital discharge. Pediatrics. 2009 May;123(5):1424-9. doi: 10.1542/peds.2009-0559. PMID 19403510
- [Background] Kakefuda I, Yamanaka T, Stallones L, Motomura Y, Nishida Y. Child restraint seat use behavior and attitude among Japanese mothers. Accid Anal Prev. 2008 May;40(3):1234-43. doi: 10.1016/j.aap.2008.01.013. Epub 2008 Feb 25. PMID 18460393
- [Background] Lennon A. A risky treat: exploring parental perceptions of the barriers to seating their children in the rear seats of passenger vehicles. Inj Prev. 2007 Apr;13(2):105-9. doi: 10.1136/ip.2006.012906. PMID 17446250